CLINICAL TRIAL: NCT03472937
Title: Outpatient Foley For Starting Induction of Labor at Term in Nulliparous Women: A Randomized-Controlled Study
Brief Title: Outpatient Foley For Starting Induction of Labor at Term in Nulliparous Women
Acronym: OFFSITE II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Elizabeth B. Ausbeck, Fellow, Maternal-Fetal Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F9999999
Record Dates: First submitted 2018-02-12; First posted 2018-03-21 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Pregnancy Related
Keywords: Mechanical cervical ripening; Transcervical catheter; Foley catheter for labor induction; Cervical ripening; Induction of labor
MeSH Terms: interventions — Cervical Ripening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpatient cervical ripening group (Active Comparator): Subjects in this arm will be seen in the outpatient setting, and if they qualify and are randomized to the inpatient (control) group, they will be admitted to labor and delivery the next day for cervical ripening with a transcervical Foley catheter.
  Interventions: Procedure: Transcervical Foley catheter placement for cervical ripening
- Outpatient cervical ripening group (Active Comparator): Subjects in this arm will undergo cervical ripening with a transcervical Foley catheter in the outpatient setting (intervention arm). The transcervical catheter will be placed in the office after confirmation of fetal well-being. They will then return the next day to be admitted to labor and delivery for induction of labor with oxytocin.
  Interventions: Procedure: Transcervical Foley catheter placement for cervical ripening

INTERVENTIONS:
Procedure: Transcervical Foley catheter placement for cervical ripening — Subjects will be randomized have cervical ripening with a transcervical Foley catheter in either the inpatient or outpatient setting.

SUMMARY:
The investigators are performing a randomized controlled trial investigating starting cervical ripening in the outpatient setting with a mechanical method, the transcervical Foley catheter. The objective of the study is to determine if outpatient compared to inpatient cervical ripening with a transcervical Foley catheter in nulliparous women undergoing induction shortens the time spent in labor and delivery (from the time of admission to the time of delivery).

DETAILED DESCRIPTION:
Approximately 20-25% of pregnant women undergo an induction of labor, and a large percentage of these women require cervical ripening in order to "ready" the cervix for induction. In the setting of an unfavorable cervix, induction of labor with oxytocin alone can be associated with longer times to delivery, uterine tachysystole (uterine contractions that are too frequent), and increased rates of cesarean delivery.

Outpatient cervical ripening is an attractive option for both women and their physicians, as this allows for the potential to spend less time in the hospital and more time in the comforts of the patient's own home.

The investigators will conduct a randomized controlled trial comparing outpatient to inpatient cervical ripening using a transcervical Foley catheter. Women will be randomized to undergo inpatient or outpatient transcervical Foley catheter cervical ripening beyond their 39th week of gestation. Women and their infants will be followed until the time of their discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Nulliparous
* Singleton gestation
* Gestational age between 39+0 and 42+0 weeks
* Vertex presentation
* Modified Bishop score <5 and cervical dilation ≤ 2 cm
* No prior cesarean or prior uterine surgery
* Resides within 30 minutes of UAB Hospital
* Access to a telephone
* Reliable transportation

Exclusion Criteria:

* Unsuitable for outpatient cervical ripening (e.g., IUGR, oligohydramnios, polyhydramnios, gestational hypertension or preeclampsia, complex maternal disease, provider discretion). Patients with well controlled Class A or B DM or chronic hypertension will be eligible.
* Latex allergy
* Contraindication to induction of labor
* Evidence of labor
* Fetal demise
* Fetal anomaly
* Inability to give consent (e.g., inability to read or write)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Total time from admission to delivery | From baseline to the time of delivery (baseline is from admission)

SECONDARY OUTCOMES:
Modified Bishop score on admission | At baseline
Evaluation of patient satisfaction with care | Within 2-4 days after delivery
  Assessed through survey adapted from "Six Simple Questions Survey," which has been published by Harvey et al (Harvey et al. Evaluation of satisfaction with midwifery care. Midwifery. 2002 Dec; 18(4):260-7.) This survey has 6 questions to assess perceptions of satisfaction with care. The questions include questions such as, "I had appropriate and adequate control over my care," "The person(s) responsible for my care are/were caring and compassionate," and "Problems that have arisen up to now have not been dealt with effectively." The scare ranges from 1-7, with 1 representing Strongly Disagree and 7 representing Strongly Agree.
Evaluation of patient experience on labor and delivery | Within 2-4 days after delivery
  Assessed through survey adapted from "Labor and Delivery Index (LADY-X" Survey, which has been published by Gartner et al (Gartner et al. Calculating Preference Weights for the Labor and Delivery Index: A Discrete Choice Experiment on Women's Birth Experiences. Value Health. 2015 Sep; 18(6):856-864.) This survey has 7 questions to assess experiences during labor and birth. Each question then has 3 answer choices that describe how good/poor the experience was. An example of a question is, "Taking your wishes seriously during childbirth." The answers then include "very seriously, sufficiently seriously, or insufficiently seriously."
Evaluation of pain experienced during childbirth | From placement of Foley bulb to delivery
  Assessed through survey that contains 4 questions. The first 3 questions assess pain (worst pain during labor, overall pain during labor, and worse pain during placement of the Foley balloon). The 4th question asks how likely a patient is to recommend her method of induction to a friend/family member. The scale ranges from 0-100, with 0 representing no pain or very unlikely and 100 representing pain as bad as it could possibly be or very likely. The patient is instructed to place a hash mark over the line.
Vaginal bleeding greater than bloody show | From placement of Foley bulb to delivery
  Vaginal bleeding that is like a period or more
Total hospital duration | From hospital admission to hospital discharge (generally less than one week)
Rates of acetaminophen use | From placement of Foley bulb to 24 hours
Rates of calls to the obstetrical triage unit | From placement of Foley bulb to 24 hours
Early admission or early visit to the obstetrical triage unit prior to scheduled induction of labor time | From placement of Foley bulb to 24 hours
Rates of spontaneous rupture of membranes between Foley bulb placement and admission | From placement of Foley bulb to 24 hours
Non-reassuring fetal heart rate tracings 30-minutes after Foley bulb placement | From placement of Foley bulb to 30 minutes
Total duration of time of neuraxial anesthesia use | From baseline to delivery
Total time of oxytocin infusion | From baseline to delivery
Maximum oxytocin rate | From baseline to delivery
Highest maternal intrapartum temperature | From baseline to delivery
Rates of chorioamnionitis | From baseline to delivery
Rates of endometritis | From delivery until 30 days post-discharge
Mode of delivery | From baseline to delivery
  Rates of vaginal delivery, cesarean delivery, and operative vaginal delivery (vacuum or forceps)
Postpartum hemorrhage | At delivery
Rates of hospital readmission within 30 days | From hospital discharge until 30 days post-discharge
Rates of 5-minute Apgar score <7 | From time of delivery up to 5 minutes post-delivery
Rates of umbilical cord artery pH <7.1 | From time of delivery up to 5 minutes post-delivery
Rates of umbilical cord artery base deficit <-12 | From time of delivery up to 5 minutes post-delivery
Rates of neonatal intensive care unit admissions | After delivery and before neonatal discharge (generally less than one week)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Ausbeck, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Background] Kelly AJ, Alfirevic Z, Ghosh A. Outpatient versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2013 Nov 12;(11):CD007372. doi: 10.1002/14651858.CD007372.pub3. PMID 24222365
- [Background] Amorosa JM, Stone JL. Outpatient cervical ripening. Semin Perinatol. 2015 Oct;39(6):488-94. doi: 10.1053/j.semperi.2015.07.014. Epub 2015 Sep 11. PMID 26365009
- [Background] O'Brien JM, Mercer BM, Cleary NT, Sibai BM. Efficacy of outpatient induction with low-dose intravaginal prostaglandin E2: a randomized, double-blind, placebo-controlled trial. Am J Obstet Gynecol. 1995 Dec;173(6):1855-9. doi: 10.1016/0002-9378(95)90440-9. PMID 8610775
- [Background] Sciscione AC, Muench M, Pollock M, Jenkins TM, Tildon-Burton J, Colmorgen GH. Transcervical Foley catheter for preinduction cervical ripening in an outpatient versus inpatient setting. Obstet Gynecol. 2001 Nov;98(5 Pt 1):751-6. doi: 10.1016/s0029-7844(01)01579-4. PMID 11704164
- [Background] McKenna DS, Costa SW, Samuels P. Prostaglandin E2 cervical ripening without subsequent induction of labor. Obstet Gynecol. 1999 Jul;94(1):11-4. doi: 10.1016/s0029-7844(99)00244-6. PMID 10389710
- [Background] Rayburn W, Gosen R, Ramadei C, Woods R, Scott J Jr. Outpatient cervical ripening with prostaglandin E2 gel in uncomplicated postdate pregnancies. Am J Obstet Gynecol. 1988 Jun;158(6 Pt 1):1417-23. doi: 10.1016/0002-9378(88)90376-6. PMID 3289398
- [Background] Sawai SK, O'Brien WF, Mastrogiannis DS, Krammer J, Mastry MG, Porter GW. Patient-administered outpatient intravaginal prostaglandin E2 suppositories in post-date pregnancies: a double-blind, randomized, placebo-controlled study. Obstet Gynecol. 1994 Nov;84(5):807-10. PMID 7936516
- [Background] Biem SR, Turnell RW, Olatunbosun O, Tauh M, Biem HJ. A randomized controlled trial of outpatient versus inpatient labour induction with vaginal controlled-release prostaglandin-E2: effectiveness and satisfaction. J Obstet Gynaecol Can. 2003 Jan;25(1):23-31. doi: 10.1016/s1701-2163(16)31079-9. PMID 12548322
- [Background] Wilkinson C, Bryce R, Adelson P, Turnbull D. A randomised controlled trial of outpatient compared with inpatient cervical ripening with prostaglandin E(2) (OPRA study). BJOG. 2015 Jan;122(1):94-104. doi: 10.1111/1471-0528.12846. Epub 2014 May 14. PMID 24824157
- [Background] Jozwiak M, Bloemenkamp KW, Kelly AJ, Mol BW, Irion O, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2012 Mar 14;(3):CD001233. doi: 10.1002/14651858.CD001233.pub2. PMID 22419277
- [Background] Dowswell T, Kelly AJ, Livio S, Norman JE, Alfirevic Z. Different methods for the induction of labour in outpatient settings. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD007701. doi: 10.1002/14651858.CD007701.pub2. PMID 20687092
- [Background] Sciscione AC, Bedder CL, Hoffman MK, Ruhstaller K, Shlossman PA. The timing of adverse events with Foley catheter preinduction cervical ripening; implications for outpatient use. Am J Perinatol. 2014 Oct;31(9):781-6. doi: 10.1055/s-0033-1359718. Epub 2013 Dec 17. PMID 24347259
- [Background] Henry A, Madan A, Reid R, Tracy SK, Austin K, Welsh A, Challis D. Outpatient Foley catheter versus inpatient prostaglandin E2 gel for induction of labour: a randomised trial. BMC Pregnancy Childbirth. 2013 Jan 29;13:25. doi: 10.1186/1471-2393-13-25. PMID 23356673
- [Derived] Alfirevic Z, Gyte GM, Nogueira Pileggi V, Plachcinski R, Osoti AO, Finucane EM. Home versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD007372. doi: 10.1002/14651858.CD007372.pub4. PMID 32852803
- [Derived] Ausbeck EB, Jauk VC, Xue Y, Files P, Kuper SG, Subramaniam A, Casey BM, Szychowski JM, Harper LM, Tita AT. Outpatient Foley Catheter for Induction of Labor in Nulliparous Women: A Randomized Controlled Trial. Obstet Gynecol. 2020 Sep;136(3):597-606. doi: 10.1097/AOG.0000000000004041. PMID 32769658
- See also: WHO Recommendations for Induction of Labour — http://apps.who.int/iris/bitstream/10665/44531/1/9789241501156_eng.pdf